CLINICAL TRIAL: NCT06902350
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of CS231295 in Subjects With Advanced Solid Tumors
Brief Title: Safety, Pharmacokinetics and Preliminary Efficacy of CS231295 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS231295-101
Record Dates: First submitted 2025-03-17; First posted 2025-03-30 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Neoplasms; Glioblastoma, Adult; Small Cell Lung Carcinoma (SCLC)
MeSH Terms: conditions — Neoplasms; Glioblastoma; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CS231295 (Experimental): two phases: dose escalation and cohort expansion. The dose escalation part is further divided into single-dose and multiple-dose administration.
  In the cohort expansion part, only multiple doses.
  Interventions: Drug: CS231295

INTERVENTIONS:
Drug: CS231295 — oral tablet. Only one dose on C0D1 in single-dose period. Once daily from C1D1 until disease progression, death, intolerable toxicity, loss to follow-up, withdrawal of informed consent, or the end of the trial, whichever occurs first, in multiple-dose period in both escalation and cohort expansion phases.

SUMMARY:
This trial is a single-arm, open-label, first-in-human study of CS231295, comprising two phases: dose escalation (including single-dose and multiple-dose) and cohort expansion. The Dose-Limiting Toxicity (DLT) observation period includes 6 days for single-dose and the first cycle (28 days) for multiple-dose. The overall study consists of screening period, treatment period, and follow-up period.

The primary objectives of this study are to evaluate the safety, tolerability and pharmacokinetic (PK) characteristics of CS231295 in patients with advanced solid tumors, and to recommended Phase 2 dose(s) (RP2D) of CS231295 in appropriate tumor(s).

ELIGIBILITY:
Inclusion Criteria:

1. Understand and sign the informed consent form voluntarily.
2. ≥18 years old when signing the informed consent, regardless of sex.
3. Have histologically or cytologically confirmed unresectable advanced, recurrent, or metastatic solid tumors (including but not limited to small cell lung cancer, glioblastoma, urothelial carcinoma, endometrial cancer, cervical cancer, ovarian cancer, breast cancer, and liver cancer) for which standard therapy has failed or was intolerable, and currently no standard treatment is available.

   * Radiological or histopathological evidence indicating disease progression should be documented.
   * Intolerance is defined as discontinuation of treatment due to adverse events during therapy.
   * Recurrence is based on radiological or histopathological results.
4. For glioblastoma: at least one measurable intracranial tumor lesion according to the RANO 2.0 criteria. For other solid tumors: at least one measurable lesion according to RECIST v1.1 criteria. Note: Target lesions can be located in previously irradiated areas, but must be confirmed by imaging to show disease progression after radiation.
5. For glioblastoma: KPS score ≥60. For other solid tumors: ECOG performance status of 0 or 1.
6. Meet the following laboratory criteria (without receiving any blood products, hematopoietic growth factors, albumin, or other treatments within 14 days prior to testing, except iron supplements):

   * Hematology: Hemoglobin (Hb) ≥100 g/L, absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet (PLT) count ≥100×10^9/L.
   * Biochemistry: 1) Dose escalation phase: Serum creatinine (Cr) ≤ upper limit of normal (ULN); total bilirubin (TBIL) ≤1.25×ULN; alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤1.5×ULN (for subjects with liver metastases or hepatocellular carcinoma: ≤3×ULN). 2) Cohort expansion phase: Cr ≤1.5×ULN; TBIL ≤1.5×ULN; ALT, AST ≤2.5×ULN (for subjects with liver metastases or hepatocellular carcinoma: ≤5×ULN).
   * Coagulation: International normalized ratio (INR) ≤1.5×ULN; prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN (for participants receiving prophylactic anticoagulation, the INR and APTT should be within a safe and effective therapeutic range as judged by the investigator).
   * Urinalysis: Urine protein <2+; if ≥2+, a 24-hour urine protein quantification should be performed. <1 g/24 h can be enrolled but ≥1 g/24 h is prohibited. without quantification when urine protein ≥2+ is not allowed.
7. Expected survival ≥12 weeks.
8. Cohort Expansion Phase: 1) Cohort 1: Histologically or cytologically confirmed small cell lung cancer (SCLC) that has progressed or recurred after at least two lines of systemic chemotherapy (including a platinum-based regimen). Note: A new line of treatment is defined as a change in treatment due to disease progression, not due to toxicity or other reasons. Re-initiation of the same treatment regimen after initial progression is considered a new line of treatment. 2) Cohort 2: Recurrent or progressive glioblastoma confirmed by histopathology or imaging, which has progressed or recurred after at least one prior treatment with temozolomide.

Exclusion Criteria:

1. Received any form of intracranial radiotherapy within 3 months prior to the first dose.
2. Received any anti-tumor treatment (including but not limited to chemotherapy, targeted therapy, immunotherapy, cellular therapy, radiation therapy [see exclusion criterion #1 for head], endocrine anti-tumor therapy, tumor embolization) or unapproved investigational drugs or devices within 28 days prior to the first dose. Also, received Traditional Chinese Medicine (TCM) approved by the National Medical Products Administration (NMPA) for treating malignant tumors within 14 days prior to the first dose.
3. Previously received Aurora kinase inhibitors.
4. Used strong inducers or inhibitors of cytochrome P450 3A (CYP3A) enzymes within 14 days prior to the first dose or are still within 7 half-lives of such drugs (whichever is longer).
5. For glioblastoma only: >5 mg/day dexamethasone or equivalent doses of other glucocorticoids for systemic treatment related to glioblastoma within 1 week prior to the first dose.
6. Underwent major surgery (cranial, thoracic, or abdominal) within 28 days prior to the first dose or have unresolved wounds, ulcers, or fractures as judged by the investigator at screening.
7. Have unresolved toxicities from previous treatments that have not recovered to CTCAE v5.0 grade ≤1, except for alopecia or laboratory abnormalities deemed no clinical significant by the investigator.
8. History of other primary malignancies within 5 years prior to the first dose, except for adequately treated in situ carcinoma, non-melanoma skin cancer, or malignant melanosis.
9. For solid tumors other than glioblastoma: Unstable brain metastases. Stable brain metastases are allowed if:

   * No immediate or planned local treatment for brain metastases during the study.
   * No neurological symptoms or signs (e.g., increased intracranial pressure, seizures, cognitive impairment) at screening.
   * Brain lesions stable for ≥2 weeks prior to the first dose without corticosteroid or anticonvulsant treatment.
10. Leptomeningeal metastasis (except glioblastoma).
11. Severe brain herniation or risk thereof.
12. For glioblastoma only: who had wafer(s) implantation during surgery.
13. Received drainage of pleural effusion, ascites, or pericardial effusion within 1 month prior to the first dose or have significant clinical symptoms (e.g., chest tightness, shortness of breath, dyspnea).
14. Uncontrolled or significant cardiovascular disease, including:

    * NYHA Class II or higher congestive heart failure, unstable angina, myocardial infarction within 6 months prior to the first dose, or arrhythmias requiring treatment, left ventricular ejection fraction (LVEF) <50% at screening.
    * Primary cardiomyopathy (e.g., dilated, hypertrophic, arrhythmogenic right ventricular, restrictive, or unclassified cardiomyopathy).
    * Symptomatic coronary artery disease requiring medication at screening.
    * Clinically significant QTcF prolongation history or QTcF >470 ms (females) and >450 ms (males) at screening.
    * Significant cerebrovascular accident (including cerebral hemorrhage, transient ischemic attack) within 6 months prior to the first dose.
    * Use of ≥3 antihypertensive drug components within 14 days prior to the first dose or inadequately controlled blood pressure (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg) at screening.
    * Other cardiovascular conditions deemed unsuitable by the investigator.
15. Poorly controlled diabetes (fasting glucose >10 mmol/L).
16. Significant gastrointestinal abnormalities at screening that may affect drug intake, transport, or absorption (e.g., inability to swallow, chronic diarrhea, bowel obstruction, small bowel resection, or total gastrectomy).
17. Clinically significant hemoptysis or tumor bleeding within 14 days prior to the first dose; significant active bleeding within 2 months prior to the first dose (e.g., gastrointestinal bleeding); currently on anticoagulants (e.g., warfarin, phenprocoumon, but low-dose aspirin and heparin for prophylaxis allowed); high-risk bleeding tendency at screening (e.g., esophageal varices, active ulcerative lesions, positive occult blood in stool, imaging evidence of tumor invasion into large vessels).
18. Serious thromboembolic events within 6 months prior to the first dose (e.g., arterial thrombosis, pulmonary embolism, deep vein thrombosis). Implanted venous port or catheter-related thrombi, superficial vein thrombi, or those deemed stable and not requiring emergency medical intervention are not considered "serious."
19. Active infection requiring intravenous treatment at screening. Severe infections (e.g., hospitalization due to infection, bacteremia, severe pneumonia complications) within 28 days prior to the first dose. Patients receiving prophylactic antibiotics (e.g., for urinary tract infections or COPD exacerbations) can be enrolled.
20. Known active tuberculosis, currently receiving anti-tuberculosis treatment, or received anti-tuberculosis treatment within 1 year prior to the first dose.
21. Active hepatitis B (HBsAg or HBcAb positive with viral replication) or hepatitis C (HCV antibody positive with viral replication) at screening.
22. Human immunodeficiency virus (HIV) infection or syphilis infection (positive specific antibody test followed by positive non-specific antibody test) at screening.
23. Allergy or hypersensitivity to any component of the trial drug or known excipients, or history of severe allergic diseases.
24. History of organ transplantation or allogeneic hematopoietic stem cell transplantation.
25. History of alcohol abuse or drug abuse.
26. Any psychiatric or cognitive disorder that may limit understanding of informed consent, compliance with the protocol, or participation in the trial.
27. Unwilling or unable to use effective contraception methods during the entire treatment period and up to 3 months after the last dose for women of childbearing potential (defined as having experienced menarche and not undergone successful artificial sterilization [hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or not postmenopausal) or male patients whose partners are women of childbearing potential; pregnant or breastfeeding women.
28. Other conditions deemed unsuitable for participation in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
incidence of dose-limiting toxicity (DLT) | 34 days after, that is 6 days after single-dose and 28 days after first administration in multiple-dose
maximum tolerated dose (MTD) | dose escalation part, about 2 years
incidence of adverse events (AEs) | from first administration to 28 days after last administration or next anti-tumor therapy, whichever occurs first
  Number of participants with AE(s)
Pharmacokinetic parameters: Time to Maximum Concentration (Tmax) | during treatment, up to 11 cycles, 28 days in one cycle
Pharmacokinetic parameters: Maximum Concentration (Cmax) | during treatment, up to 11 cycles, 28 days in one cycle
Pharmacokinetic parameters: Area Under the Concentration-time Curve(AUC) | during treatment, up to 11 cycles, 28 days in one cycle
Pharmacokinetic parameters: Trough Concentration (Ctrough) | during treatment, up to 11 cycles, 28 days in one cycle
Pharmacokinetic parameters: Accumulation Ratio (Rac) | during treatment, up to 11 cycles, 28 days in one cycle
Pharmacokinetic parameters: Elimination Half-life (t1/2) | during treatment, up to 11 cycles, 28 days in one cycle
Pharmacokinetic parameters: Clearance over Fractional Bioavailability (CL/F) | during treatment, up to 11 cycles, 28 days in one cycle
Pharmacokinetic parameters: Volume of Distribution at Steady State over Fractional Bioavailability (Vz/F) | during treatment, up to 11 cycles, 28 days in one cycle

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | during study, expected average one year
Disease control rate (DCR) | during study, expected average one year
Duration of Response (DOR) | during study, expected average one year
Time to Progression (TTP) | during study, expected average one year
Time to Response (TTR) | during study, expected average one year
progression-free survival (PFS) | during study, expected average one year
Overall Survival (OS) | during study, expected average one year

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, M.D., Principal Investigator — Beijing Tiantan Hospital; Ying Cheng, M.D., Principal Investigator — Jilin Provincial Tumor Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Jilin Cancer Hospital, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No